CLINICAL TRIAL: NCT07316777
Title: Protocol for Development and Implementation of the Saudi CABG Audit and Registry: A Prospective National Clinical Registry
Brief Title: Saudi CABG Audit and Registry
Acronym: SCAR
Status: Not yet recruiting | Type: Observational
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Uthman Aluthman, Consultant Cardiac Surgeon, King Faisal Specialist Hospital & Research Center
Other Study IDs: 2251502
Record Dates: First submitted 2025-11-27; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Bypass Graft (CABG)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prospective Clinical Data Collection — The intervention consists of systematic, prospective collection of standardized clinical, operative, and follow-up data for all adult patients undergoing coronary artery bypass grafting (CABG) at participating centers. Data are recorded across predefined time points, including preoperative assessment, intraoperative details, postoperative in-hospital outcomes, and follow-up at 30 days, 3 months, 6 months, and 1 year. Variables include demographics, comorbidities, cardiac status, operative technique, complications, readmissions, mortality, and patient-reported quality-of-life measures (EQ-5D and SF-36). No treatments are assigned. The registry functions solely as an observational platform for quality improvement, benchmarking, and long-term outcome monitoring.

SUMMARY:
The Saudi CABG Audit and Registry (SCAR) is a prospective, multicenter national clinical quality registry designed to systematically collect perioperative and long-term outcome data for all patients undergoing coronary artery bypass grafting (CABG) in Saudi Arabia. The registry will begin with a pilot phase in selected tertiary cardiac centers and will progressively expand to national coverage. SCAR captures detailed information on patient demographics, cardiac status, operative techniques, postoperative outcomes, and 1-year follow-up, including patient-reported quality-of-life measures (EQ-5D and SF-36). The aim is to establish a standardized national platform for benchmarking, quality improvement, and real-world evidence generation to support clinical decision-making and health policy development in cardiac surgery. Data are collected prospectively through secure electronic systems, anonymized before central storage, and analyzed using standardized definitions aligned with international registries such as STS and E-CABG.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older
* Undergoing isolated CABG
* Undergoing CABG with concomitant procedures (e.g., valve repair or replacement)
* Undergoing on-pump, off-pump, minimally invasive, or robotic CABG
* Procedures performed electively, urgently, or emergently

Exclusion Criteria:

* Redo CABG when the primary operative record is not available
* Patients younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) undergoing coronary artery bypass grafting (CABG) at participating cardiac surgery centers in Saudi Arabia. The population includes individuals receiving isolated CABG or CABG with concomitant procedures, performed electively, urgently, or emergently, using on-pump, off-pump, minimally invasive, or robotic approaches.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of In-hospital mortality | From date of surgery through hospital discharge, an average of 7-10 days.
  In-hospital all-cause mortality following coronary artery bypass grafting (CABG), recorded from the time of surgery until discharge. Mortality will be determined using standardized definitions aligned with major cardiac surgery registries such as STS and E-CABG.
Incidence of 30-day major adverse cardiac and cerebrovascular events (MACCE) | 30 days post-surgery
  Composite endpoint including 30-day all-cause mortality, stroke, and myocardial infarction after coronary artery bypass grafting (CABG). Event definitions follow standardized criteria used in major cardiac surgery registries, including STS and E-CABG.
Incidence of Deep sternal wound infection (DSWI) | From surgery until 30 days post-operation
  Incidence of deep sternal wound infection following coronary artery bypass grafting (CABG), defined according to Centers for Disease Control and Prevention (CDC) criteria. Includes infections involving muscle, bone, or mediastinum requiring surgical intervention, antibiotics, or drainage.
Unplanned reoperation for bleeding, tamponade, or graft-related technical failure | Perioperative/Periprocedural
  Incidence of unplanned return to the operating room after coronary artery bypass grafting (CABG) due to postoperative bleeding, cardiac tamponade, or graft-related technical failure. Events follow standardized definitions aligned with international cardiac surgery registries.

SECONDARY OUTCOMES:
Intensive care unit (ICU) length of stay | From the date of surgery through initial ICU discharge (average of 3-5 days).
  Duration of postoperative stay in the intensive care unit following CABG surgery, measured in hours or days. Includes all ICU readmissions during the index hospitalization.
Total hospital length of stay | From the date of surgery through hospital discharge (average of 7-10 days).
  Duration of hospitalization from the day of surgery until discharge, measured in days. Includes all in-hospital recovery time after CABG.
Duration of mechanical ventilation | From completion of surgery through extubation, an average of 12-24 hours
  Total time on postoperative mechanical ventilation following CABG surgery, measured in hours. Includes any episodes of re-intubation requiring ventilatory support.
Incidence of 30-day readmission | Within 30 days post-discharge
  Incidence of all-cause hospital readmission occurring within 30 days of discharge after CABG surgery.
Number of Participants with Post Operative Acute kidney injury (AKI) | From date of surgery through hospital discharge, an average of 7-10 days.
  Occurrence of acute kidney injury following CABG, defined according to KDIGO criteria (increase in serum creatinine ≥0.3 mg/dL within 48 hours, ≥1.5× baseline within 7 days, or urine output <0.5 mL/kg/h for 6 hours).
Incidence of New renal replacement therapy Initiation | From date of surgery through hospital discharge, an average of 7-10 days.
  Initiation of postoperative renal replacement therapy (intermittent dialysis or continuous renal replacement therapy) that was not required preoperatively.
Number of Participants with post operative New-onset atrial fibrillation | From date of surgery through hospital discharge, an average of 7-10 days.
  Incidence of atrial fibrillation requiring medical or procedural intervention following CABG, documented on electrocardiography or continuous telemetry.
Blood product utilization | Intraoperative through 24 hours post-surgery
  Number and type of transfused blood products (red blood cells, plasma, platelets, cryoprecipitate) during and after CABG surgery.
One-year survival | 1 year post-surgery
  All-cause survival at 1 year following CABG surgery, assessed through clinical follow-up and health records.
One-year MACCE | 1 year post-surgery
  Composite of all-cause mortality, stroke, myocardial infarction, and repeat revascularization occurring within 1 year after CABG.
Return to work or usual activity | 1 year post-surgery
  Proportion of patients who resume employment or routine daily activity within 1 year after CABG.
EuroQol-5 Dimension (EQ-5D) | Baseline, 6 months, 1 year
  Change in health-related quality of life after coronary artery bypass grafting (CABG), measured using the EuroQol 5-Dimension (EQ-5D) questionnaire. The EQ-5D index score ranges from 0 to 1, where 0 represents the worst possible health state and 1 represents the best possible health state. Higher scores indicate better health-related quality of life. The EQ-5D will be administered at baseline, 6 months, and 1 year to evaluate changes over time.
Short Form Health Survey (SF-36) | Baseline, 6 months, and 1 year post-surgery
  Change in health-related quality of life after coronary artery bypass grafting (CABG), measured using the 36-Item Short Form Health Survey (SF-36). Each of the eight domains is scored from 0 to 100, where 0 represents the worst health status and 100 represents the best health status. Higher scores indicate better functional and mental health outcomes. The SF-36 will be administered at baseline, 6 months, and 1 year to assess longitudinal recovery.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alpert JS. Are data from clinical registries of any value? Eur Heart J. 2000 Sep;21(17):1399-401. doi: 10.1053/euhj.2000.2265. No abstract available. PMID 10952831
- [Background] Wyse RK, Taylor KM. The development of an international surgical registry: the ECSUR project. The European Cardiac Surgical Registry. Eur J Cardiothorac Surg. 1999 Jul;16(1):2-8. doi: 10.1016/s1010-7940(99)00129-3. PMID 10456394
- [Background] Bridgewater B; Society for Cardiothoracic Surgery in GB and Ireland. Cardiac registers: the adult cardiac surgery register. Heart. 2010 Sep;96(18):1441-3. doi: 10.1136/hrt.2010.194019. Epub 2010 May 29. PMID 20511631
- [Background] Gitt AK, Bueno H, Danchin N, Fox K, Hochadel M, Kearney P, Maggioni AP, Opolski G, Seabra-Gomes R, Weidinger F. The role of cardiac registries in evidence-based medicine. Eur Heart J. 2010 Mar;31(5):525-9. doi: 10.1093/eurheartj/ehp596. Epub 2010 Jan 20. No abstract available. PMID 20093258
- [Background] Biancari F, Ruggieri VG, Perrotti A, Svenarud P, Dalen M, Onorati F, Faggian G, Santarpino G, Maselli D, Dominici C, Nardella S, Musumeci F, Gherli R, Mariscalco G, Masala N, Rubino AS, Mignosa C, De Feo M, Della Corte A, Bancone C, Chocron S, Gatti G, Gherli T, Kinnunen EM, Juvonen T. European Multicenter Study on Coronary Artery Bypass Grafting (E-CABG registry): Study Protocol for a Prospective Clinical Registry and Proposal of Classification of Postoperative Complications. J Cardiothorac Surg. 2015 Jun 30;10:90. doi: 10.1186/s13019-015-0292-z. PMID 26123033